CLINICAL TRIAL: NCT03222232
Title: Catheter-related Bloodstream Infections in Patients With Intestinal Failure Receiving Home Parenteral Support: Risks Related to a Catheter-salvage-strategy.
Brief Title: Catheter Salvage in Intestinal Failure Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Palle Bekker Jeppesen, Professor, MD, Rigshospitalet, Denmark
Other Study IDs: CVC salvage study
Record Dates: First submitted 2017-07-16; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Intestinal Failure; Catheter-Related Bloodstream Infection (CRBSI) Nos
Keywords: intestinal failure; catheter-related bloodstream infections; catheter salvage; recurrent infections; home parenteral support
MeSH Terms: conditions — Intestinal Failure; Pyloric Stenosis, Hypertrophic; Reinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic intestinal failure patients: Patients with chronic intestinal failure on home parenteral support and enrolled in the Copenhagen Intestinal failure database between January 1, 2002 and December 31, 2015.
  Interventions: Behavioral: catheter salvage

INTERVENTIONS:
Behavioral: catheter salvage — In each case of catheter-related bloodstream infection the management of the central venous catheter was registred to evaluate the future risk of new infections

SUMMARY:
This is an observational study evaluating a catheter salvage strategy in relation to catheter-related bloodstream infections in patients with chronic intestinal failure dependent on home parenteral support. The study is confined to the period 2002 to 2016.

DETAILED DESCRIPTION:
In chronic intestinal failure patients receiving home parenteral support (HPS), catheter-related bloodstream infections (CRBSIs) frequently results in replacement of their tunneled central venous catheters (CVCs) which may lead to future loss of central venous access.

This observational study investigates the consequences of a catheter-salvage-strategy related to CRBSIs according to different causative microorganisms, and short- and long-term risk of recurrence of the CRBSI. The study is based on the Copenhagen Intestinal failure database, which is a web-based database with retrospective data collection performed by reviews of medical charts from all adult intestinal failure patients discharged with home parenteral support from the Department of Medical Gastroenterology, Rigshospitalet.

ELIGIBILITY:
Inclusion Criteria:

* chronic intestinal failure dependent on home parenteral support and enrolled in the Copenhagen Intestinal failure database

Exclusion Criteria:

* Never discharged on home parenteral support

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with intestinal failure, characterised by a reduction in the guts capacity to absorb macronutrients and/or fluid and electrolytes below what is necessary to maintain health, and therefore parenteral support (nutrition and/or fluids and electrolytes) is required to sustain life. Patient initiated on Home parenteral support was entered into the Copenhagen Intestinal failure database, and thereby eligible in this cohorte study.
Sampling Method: Non-Probability Sample
Enrollment: 715 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
new catheter-related bloodstream infections | 2002 to 2016
  The occurrence of catheter-related bloodstream infection after either catheter salvaged (retained central venous catheter) or replaced central venous catheter (new central venous catheter)

SECONDARY OUTCOMES:
recurrent catheter-related bloodstream infections | 2002 to 2016
  A recurrent infection was defined as a CRBSI with identical microorganism and antibiogram occurring within 100 days of the previous CRBSI in a salvaged CVC.
relapse catheter-related bloodstream infection | 2002 to 2016
  A relapse infection was defined as recrudescence of the same causative microorganisms with identical antibiogram within 30 days of the previous CRBSI in a salvaged CVC.
primary salvage rate | 2002 to 2016
  The primary salvage rate was defined by the CVC status at hospital discharge. Because of the database setup and retrospective design of the study, all cases were included regardless of main reason to CVC removal (e.g. septic shock, severe sepsis, concomitant CVC problems and secondary or metastatic complications).

CONTACTS AND LOCATIONS:
Overall Officials: Siri Tribler, MD, Principal Investigator — Department of Medical gastroenterology, Rigshospitalet
Locations (1):
- Rigshospitalet, abdominalcentret, Medicinsk Gastroenterologisk klinik CA, 2121, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No